CLINICAL TRIAL: NCT04725708
Title: The Effect of Intraoperative Arterial Oxygen Levels on Cognitive Functions After Coronary Bypass Graft Surgery
Brief Title: Cognitive Functions on Coronary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tugba Onur, Principal investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bursa YIERH
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Neurocognitive Disorders
Keywords: cardiovascular surgery; cerebral oxymetre; neurocognitive assessment
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normoxy (Experimental): Group 1(n=50) FiO2%40, PaO2<180 ve PaO2≥80mmHg MMSE will be applied to patients before surgery. At the determined measurement times body and blood temperature, SpO2, HR, MAP, PH, blood gas lactate, blood gas base deficit, urine output, PaO2, PaCO2, Htc, FiO2, right and left rSO2 values were monitored.
  An rSO2 less than 45% triggered an alarm, the anesthesiologist timed the event, and after 60 seconds initiated an intervention protocol means; PaO2 levels were checked, PaO2> 100 mmHg was achieved, if not improved, pump blood flow, mean arterial pressure were increased, if there is still no response and hematocrit <20%, patients were scheduled for erythrocyte transfusion until the rSO2 was restored to at least 60% at both probes.In the postoperative period, at the 24th hour, when routine cardiological controls were performed 1., 3., 6. Simultaneous MMSE will be repeated in months.
  Interventions: Procedure: procedure: cerebral oxygenation intervention
- hyperoxia (Experimental): Group 2(n=50) FiO2%100, PaO2≥180mmHg MMSE will be applied to patients before surgery. At the determined measurement times body and blood temperature, SpO2, HR, MAP, PH, blood gas lactate, blood gas base deficit, urine output, PaO2, PaCO2, Htc, FiO2, right and left rSO2 values were monitored..In the postoperative period, at the 24th hour, when routine cardiological controls were performed 1., 3., 6. Simultaneous MMSE will be repeated in months.
  Interventions: Procedure: procedure: cerebral oxygenation intervention

INTERVENTIONS:
Procedure: procedure: cerebral oxygenation intervention — During the surgery, cerebral oxygenation will be followed and intervention will be made to pH, PaO2, PaCO2, mean arterial pressure, hematocrit when necessary. In addition perfusion flow was maintained at or close to between 2.2-2.5 L/min/m2 . Perfusion pressure was adjusted using a phenylephrine infusion to maintain a mean arterial pressure of 50 to 70 mm Hg.

SUMMARY:
The aim of this study is to examine the effects of different but safe levels of arterial oxygen levels used in cardiac surgeries on cerebral oxygenation during the operation. It is also to investigate the effect on cognitive functions in the postoperative period. For our study the investigators will conduct a randomized control trial. Patients will be randomly assigned to one of two possible study groups according to the arterial oxygen levels.If there is any abnormality in cerebral oxygen levels during surgery, necessary intervention will be made by doctors.

DETAILED DESCRIPTION:
In most cardiovascular surgeries, patients are frequently followed up at hyperoxemic level for safety purposes against the risk of tissue hypoxia that may develop during surgery due to CPB use. At the level of hyperoxemia, there are opinions that the ischemia-reperfusion damage increases with the follow-up of CABG surgery, microcirculation is impaired and tissue oxygenation is impaired due to the resulting hyperoxemic vasoconstriction. Recent research has focused on evaluating optimal oxygen levels in CPB during cardiac surgery. However, the potential of tightly regulated intraoperative normoxia to improve POCD following cardiac surgery has not been studied prospectively.

The purpose of this study is to determine whether patients who underwent CPB and CABG, which were preserved under normoxic conditions during the intraoperative period, would have a lower incidence of early and late POCD than those exposed to hyperoxia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled to undergo elective cardiopulmonary bypass graft surgery

Exclusion Criteria:

* severe preoperative cognitive impairment(i.e. dementia, intellectual disorder)
* Non-Turkish speaking patients
* presence of end-stage organ failure
* patients requiring emergency coronary surgery
* surgical procedures requiring single lung ventilation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative neurocognitive function | 12 hours after surgery
  Change on MMSE is important for neurocognitive disorder.The MMSE consists of cognitive functions of orientation, attention, calculation, memory and language.
postoperative neurocognitive function | 24 hours after surgery
  Change on MMSE is important for neurocognitive disorder.The MMSE consists of cognitive functions of orientation, attention, calculation, memory and language.
postoperative neurocognitive function | 1 month after surgery
  Change on MMSE is important for neurocognitive disorder.The MMSE consists of cognitive functions of orientation, attention, calculation, memory and language.
postoperative neurocognitive function | 3 months after surgery
  Change on MMSE is important for neurocognitive disorder.The MMSE consists of cognitive functions of orientation, attention, calculation, memory and language.
postoperative neurocognitive function | 6 months after surgery
  Change on MMSE is important for neurocognitive disorder.The MMSE consists of cognitive functions of orientation, attention, calculation, memory and language.

SECONDARY OUTCOMES:
Extubation time after surgery | During the hospitalization for postoperative recovery ,average 8 days
  Weaning times from mechanical ventilation among patients who are followed up with the same intensive care approach after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba T ONUR, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Ümran Ü KARACA, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Filiz F ATA, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Halil Erkan H SAYAN, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Anıl A ONUR, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Canan C YILMAZ, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Ayşe Neslihan AN BALKAYA, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Cüneyt C ERİŞ, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa YIERH, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No